CLINICAL TRIAL: NCT06692023
Title: Impact of High-Intensity-NIV Vs Low-intensity-NIV on Subjective Tolerance Amomg Patients with AECOPD : a Randomised Cross-over Pilot Study
Brief Title: Impact of HI-NPPV Vs LI-NPPV on Tolerance Among AECOPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BeijingCYH-ICU-008
Record Dates: First submitted 2024-10-22; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity NPPV (Experimental): Patients will receive high-intensity NPPV
  Interventions: Device: High-intensity NPPV; Device: Low-intensity NPPV
- Low-intensity NPPV (Active Comparator): Patients will receive low-intensity NPPV
  Interventions: Device: High-intensity NPPV; Device: Low-intensity NPPV

INTERVENTIONS:
Device: High-intensity NPPV — In the high-intensity NPPV group, IPAP is initially adjusted in increments/decrements of 1-2 cmH2O, typically ranging from 20 to 30 cmH2O (or a tolerated maximum), to obtain a VT 10-15 mL/kg PBW and a respiratory rate <25 breaths/min. Subsequent adjustments to IPAP are based on the results of arterial blood gases (ABGs; up to 30 cmH2O) to achieve normocapnia (if possible), or to maximally decrease PaCO2 toward normocapnia if normocapnia can not be achieved. If PaCO2 decreases to less than 35 mmHg, IPAP will be decreased to achieve normocapnia.
Device: Low-intensity NPPV — In the low-intensity NPPV group, as well as during the 6-hour trial of low-intensity NPPV, IPAP is initially adjusted in increments/decrements of 1-2 cmH2O (up to 20 cmH2O), according to patients' tolerance, to obtain a VT 6-10 mL/kg PBW and a respiratory rate <25 breaths/min. Subsequent adjustments to IPAP are based on the results of ABGs (up to 20 cmH2O) to achieve a pH of ≥7.35 and to reduce PaCO2 to a level deemed appropriate by the attending physician.

SUMMARY:
To determine whether high-intensity NPPV, compared with low-intensity NPPV, could have an effect on the subjective tolerance in patients with an AECOPD and hypercapnia.

DETAILED DESCRIPTION:
To evaluate the subjective tolerance of high-intensity NPPV and low-intensity NPPV patients in a conscious state by two questionnaire surveys; To assess tolerance of high-intensity NPPV and low-intensity NPPV patients patient in sleeping status by PSG monitoring.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD confirmed by the 2019 criteria of the Global Initiative for Chronic Obstructive Lung Disease (GOLD);
* Arterial pH <7.35 and PaCO2 >45 mmHg at screening entry;
* PaCO2 >45 mmHg after a 6-hour trial of low-intensity NPPV.

Exclusion Criteria:

* Age <18 years
* Excessive respiratory secretions with weak cough
* Upper airway obstruction
* Recent oral, facial, or cranial trauma or surgery
* Recent gastric or esophageal surgery
* Presence of restrictive ventilatory dysfunction (eg, consolidation or removal of at least one pulmonary lobe, massive pleural effusion, chest wall deformity, continuous strapping with thoracic or abdominal bandage, or severe abdominal distension)
* Active upper gastrointestinal bleeding
* Cardiac or respiratory arrest
* Arterial oxygen tension/fraction of inspired oxygen (PaO2/FiO2) <100 mmHg
* Pneumothorax
* Obvious emphysematous bullae confirmed by chest CT scan
* Ventricular arrhythmia or myocardial ischemia
* Severe hemodynamic instability (mean arterial pressure <65 mmHg)
* Severe metabolic acidosis (pH <7.20 and bicarbonate <22 mmol/L)
* Refusal to receive NPPV or give informed consent
* Prior endotracheal intubation or tracheostomy during the current hospitalization
* A do-not-intubate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
NPPV subjective tolerance | From randomization to 2 days after randomization
  NPPV subjective tolerance is mainly evaluated through two questionnaire surveys. Questionnaire survey 1 includes 19 questions, including bloating , appetite, thirst, dryness of the mouth and nose, conjunctivitis, facial tenderness, fear, airflow shock, mask tolerance, ear pain, noise, overall tolerance of NPPV, willingness to use NPPV, confidence of using NPPV, breathless relief score, sleep quality, drowsiness in day, physical strength, and mood. Questionnaire survey 2 mainly evaluates patients' feelings of using NPPV under different emotional states, feelings of using NPPV under different physical states, and feelings of using NPPV in daily life states. Each question is scored from 0 to 100 points. The higher scores indicate better positive feedback.

SECONDARY OUTCOMES:
Effects of NPPV on sleep quality | From randomization to 2 days after randomization
  The sleep quality is assessed by PSG during night

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No